CLINICAL TRIAL: NCT05165134
Title: Influence of Short-Term Conservative Treatment Using Kinesiotape on Hallux Valgus Angle
Brief Title: Hallux Valgus Conservative Treatment
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohammed Moustafa, assistant Professor of physical therapy, University of Jazan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JU
Record Dates: First submitted 2021-12-05; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Pretest and posttest Control group randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental kinesiotape group A (Experimental): Kinesiotape group
  Interventions: Other: Kinesiotape
- Placebo kinesiotape group B (Placebo Comparator): Control group
  Interventions: Other: Kinesiotape

INTERVENTIONS:
Other: Kinesiotape — Elastic tape used for mechanical correction of the deformity in study group and placebo in control group

SUMMARY:
Studying the effect of kinesiotape on hallux valgus angle and pain in hallux valgus patients.

DETAILED DESCRIPTION:
30 patients (male and female) suffering from bilateral Halux valgus. Divided randomly into 2 groups

1. st group receive kinesiotape bilaterally for correction : Hallux valgus angle (HVA) was measured using Xray and pain was measured using VAS before applying tape and after 8 weeks of tape application.
2. nd group receive placebo tape bilaterally and had the same measurements.

2 groups were on a group of exercises

ELIGIBILITY:
Inclusion Criteria:

* mobile hallux valgus

Exclusion Criteria:

* using orthotics
* knee malalignment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Hallux valgus angle (HVA ) | 8 weeks
  Hallux valgus angle measured by x ray
Pain on metatarsophalangeal joint measured by visual analogue scale (VAS) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Ahmed, Principal Investigator — Assistant Professor of physical therapy
Locations (1):
- Jazan University, Jizan, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All will be accessible on request
Supporting Information: Study Protocol
Time Frame: March 2022
Access Criteria: Thru e mail